CLINICAL TRIAL: NCT06842212
Title: Targeted Balance Training During The Menstrual Cycle To Enhance Stability And Athletic Performance: A Randomized Controlled Trial
Brief Title: Balance Training To Enhance Stability And Athletic Performance During The Menstrual Cycle
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005603
Record Dates: First submitted 2025-01-23; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Menstrual Cycle Phase; Athletic Performance; Balance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Training (Experimental)
  Interventions: Device: Balance Training
- control group (No Intervention)

INTERVENTIONS:
Device: Balance Training — balance training exercises performed on the biodex balance system 3 sessions every week for 12 weeks
  Arms: Balance Training

SUMMARY:
This study was done to investigate the effect of balance training on improving balance and athletic performance during menstrual cycle in young athletic females Does balance training improve balance and athletic performance during the menstrual cycle? 60 athletic females will participate in the study. They will be randomly assigned into two groups. Group A will receive balance training on biodex, while group B will be the control group.

ELIGIBILITY:
Inclusion Criteria:

* Their age will be ranged from 18 to 22. Their BMI will be from 18.5 to 25 kg/cm2 - Athletes

Exclusion Criteria:

* free of musculoskeletal or neurological diseases that could affect balance/ taking any medications that affect sex hormones

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Menstrual Cycle, young Athletes
Enrollment: 60 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-02-09 (Actual); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Balance | 12 weeks
  biodex balance system device to measure balance Anterior posterior Stability index (APSI) This index is calculated using the degree of oscillation of the platform, in which low values indicated that the individual had good stability.

SECONDARY OUTCOMES:
atheletic performance | 12 weeks
  atheletic subjective performance scale
  * asking participants to rate their performance during the past week according to their own opinion.
  * Use the scale between 1-10: 1="not at all satisfied", 10="fully satisfied":
Athletic dynamic balance | 12 weeks
  Star excursion balance test (SEBT) measure the ability to maintain single leg stance on one leg while reaching as far as possible with the contralateral leg in 8 different directions, When the person demonstrates a significantly decreased reach while standing on the injured limb compared to standing on the healthy limb, the Star Excursion Balance Test has highlighted her loss of dynamic postural control

CONTACTS AND LOCATIONS:
Locations (1):
- British University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/